CLINICAL TRIAL: NCT04914104
Title: Accessible Support in Surgical Training During a Pandemic Study
Acronym: ASSIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Mark Rockley, Co-Investigtor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20210097-01H
Record Dates: First submitted 2021-05-26; First posted 2021-06-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Stress; Burnout, Professional; Depression, Anxiety
MeSH Terms: conditions — Burnout, Professional; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive free access to the mobile app Headspace and directed to access the app three times a week for at least 15 minutes.
  Interventions: Behavioral: Mindfulness Training - Headspace App
- Control (No Intervention): The control group will receive standard of care, which does not involve routine in-person or free access to mobile mindfulness therapy.

INTERVENTIONS:
Behavioral: Mindfulness Training - Headspace App — The intervention group will receive free access to the mobile app Headspace and directed to access the app three times a week for at least 15 minutes.
  Arms: Intervention

SUMMARY:
The COVID-19 pandemic has fundamentally changed the surgical trainee experience by exacerbating the difficulty of this notoriously stressful training, while limiting access to traditional avenues of mental health support. The investigators propose the application of a mobile app-based mindfulness program to address stress and burnout in the surgical training.

The proposed study is a prospective randomized, observer-blinded study including surgical trainees at the University of Ottawa in their first and second years of training. The intervention group will receive free access to the mobile app Headspace and will be encouraged to access the app three times a week for 15 minutes.

DETAILED DESCRIPTION:
The COVID-19 pandemic has fundamentally changed the surgical trainee experience. The personal risks and uncertainties of this environment have compounded the difficulty of this notoriously stressful training. Burnout in the medical profession is prolific, and health care workers are not immune to the adverse mental health effects of the pandemic. Of all health professionals, surgical trainees frequently report the highest rates of burnout and severe stress. In particular, high burnout is associated with profoundly increased rates of depression and suicidal ideation in these trainees. In addition to the adverse effects of burnout and stress on the mental health wellbeing of trainees, excessive stress in the operating room can threaten patient safety and slow motor skill acquisition.

In response, many organizations have sought out methods to mitigate the negative mental health effects of surgical training. One promising intervention is mindfulness-based stress reduction. The perception of stress in surgical trainees is mediated by both cognitive and behavioural factors, which demonstrates an opportunity for mindfulness-based stress reduction (MBSR) interventions to modulate the perceived stress. In-person MBSR has been investigated in previous randomized trials of first year surgical residents. These pilot reports describe promising feasibility and adherence to mindfulness practice, with improved stress and cognitive control in the interventional arms.

Mindfulness techniques lend themselves to self-guided instruction provided by mobile apps and are a widely available resource. Mobile app-based mindfulness practice demonstrates comparable improvements in self-reported well-being when compared with in-person mindfulness sessions. When time is a scarce commodity, participant adherence is crucial to the effectiveness of any intervention. Mindfulness-based interventions have typically boasted strong adherence exceeding an average of 16 minutes per day after 3 months, particularly when self-directed. Specifically, adherence to optional online mindfulness-based practice is promising in medical trainees, with over half of trainees voluntarily adhering to regularly scheduled online mindfulness meditation after 8 weeks. In Canadian medical students, a pilot study demonstrated improved self-compassion from mindfulness-based interventions with an average adherence of only 20 minutes per week. When compared with a traditional weekly 8-session intensive mindfulness program, an abbreviated 4-session program demonstrated comparable improvements in perceived stress and empathy.

Ironically during a pandemic when stress levels at their highest, traditional wellness programs such as in-person counselling are not available due to the social distancing protocols. The investigators propose mindfulness-based therapy in the form of a mobile app to fill this void in high risk health professionals. This study investigates the effectiveness of mindfulness therapy delivered by a mobile app in surgical residents to reduce burnout and associated repercussions during the COVID-19 pandemic.

The primary objective of this investigation is to determine if access to mindfulness therapy delivered by a mobile app is effective in improving the mental well-being in surgical trainees, when compared with the current standard of care. Mental well-being encompasses a variety of factors including stress, burnout, depression and anxiety. Additional secondary objectives include adherence to mindfulness therapy and subject satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* First and second year surgical residents
* Enrolled in the Surgical Foundations program at the University of Ottawa

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Stress | 6 weeks
  Perceived Stress Questionnaire (PSQ) (0 - 40, where low is better)
Stress | 12 weeks
  Perceived Stress Questionnaire (PSQ) (0 - 40, where low is better)
Stress | 18 weeks
  Perceived Stress Questionnaire (PSQ) (0 - 40, where low is better)
Burnout | 6 weeks
  Maslach Burnout Inventory - HSS-For Medical Personnel (MBI) (0 to 6)
Burnout | 12 weeks
  Maslach Burnout Inventory - HSS-For Medical Personnel (MBI) (0 to 6)
Burnout | 18 weeks
  Maslach Burnout Inventory - HSS-For Medical Personnel (MBI) (0 to 6)
Anxiety | 6 weeks
  DASS-21 (Depression, Anxiety and Stress Scale) (0 to 63, where low is better)
Anxiety | 12 weeks
  DASS-21 (Depression, Anxiety and Stress Scale) (0 to 63, where low is better)
Anxiety | 18 weeks
  DASS-21 (Depression, Anxiety and Stress Scale) (0 to 63, where low is better)

SECONDARY OUTCOMES:
Adherence | 6 weeks
  App usage (minutes / week)
Adherence | 12 weeks
  App usage (minutes / week)
Satisfaction with App Usage | 6 weeks
  Likhert Scale (0 to 5, where higher is better)
Satisfaction with App Usage | 12 weeks
  Likhert Scale (0 to 5, where higher is better)

IPD SHARING:
Plan to Share IPD: No